CLINICAL TRIAL: NCT02774512
Title: Phase 0 Study Aiming at Identifying Predictive Biomarkers of Biological Activity and Efficacy of Nilotinib on ZAK Target in Non-metastatic Colon Cancer
Brief Title: Predictive Biomarkers of Biological Activity and Efficacy of Nilotinib on ZAK Target in Non-metastatic Colon Cancer
Acronym: ZAK-0
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: none participant has been enrolled and recruited during the first year after competent autority autorisation.
Sponsor: Institut Bergonié (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IB 2015-03
Record Dates: First submitted 2016-04-27; First posted 2016-05-17 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib (Experimental): A specific colonoscopy is performed in order to take biopsy for biological studies to determine the ZAK-0 expression status. Then the patient receives nilotinib orally at the dose of 800 mg/day (400 mg twice a day) for 7 days. The patient is scheduled for surgery the morning after the last take of the nilotinib (12 hours). When the colectomy is performed, the surgeon collects different tumoral samples which are immediately delivered to the laboratory.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Each patient will receive nilotinib 800 mg/day every day for 7 days. Study treatment will be taken twice a day (400 mg - 2 capsules) by oral route with an interval of approximately 12 hours between two doses and should not be taken with food. The entire capsule should be swallowed with water. No food should be consumed for 2 hours before taking the drug and for at least 1 hour after it.

SUMMARY:
This is a monocentric prospective non randomized phase 0 clinical trial targeting patients with colon cancer for whom an upfront surgery has been advised by the pluridisciplinary team.

DETAILED DESCRIPTION:
This is a monocentric prospective non randomized phase 0 clinical trial targeting patients with colon cancer for whom an upfront surgery has been advised by the pluridisciplinary team. The surgical management should not be changed or delayed. The patient is seen in consultation by one of the two surgeons. The patient receives information and consents to participate to the study. A specific colonoscopy is performed in order to take biopsy for biological studies. According to the expression level of ZAK-0, the patient is included in the corresponding arm: ZAK-0 expressor or ZAK-0 non-expressor. Then the patient receives nilotinib orally at the dose of 800 mg/day (400 mg twice a day) for 7 days. The patient is scheduled for surgery the morning after the last take of the nilotinib (12 hours). When the colectomy is performed, the surgeon collects different tumoral samples which are immediately delivered to the laboratory. There are no additional changes in the clinical follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed prior any study-related procedures.
2. Histological diagnosis of colon cancer.
3. Performance status ECOG 0, 1, or 2.
4. Physical status score ASA 1 or 2.
5. Patient without metastasis.
6. No previous anti-cancer treatment for colon cancer.
7. Age ≥ 18.
8. Preoperative imaging: thorax-abdominal-pelvis CT scan within 2 months.
9. Colonoscopy and biopsies to determine ZAK-0 expression level.
10. Scheduled beginning of the treatment 7 days before surgical procedure.
11. Adequate end organ function as defined by:

    11.1. total bilirubin < 1.5 x ULN,1 11.2. SGOT and SGPT < 2.5 x ULN, 11.3. creatinine < 1.5 x ULN, 11.4. Serum amylase and lipase ≤ 1.5 x ULN, 11.5. Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related.
12. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days before initiation of study drug. Women of child-bearing potential must agree to use adequate contraception, according to investigator's instructions.

    Effective contraception must be in place :
    * During the treatment with nilotinib
    * Until 2 weeks after the end of treatment.
13. Patients must have the following laboratory values (≥ LLN (lower limit of normal) or corrected to within normal limits with supplements prior to the first dose of study medication): 13.1. Potassium ≥ LLN, 13.2. Magnesium ≥ LLN, 13.3. Phosphorus, ≥ LLN, 13.4. Total calcium (corrected for serum albumin) ≥ LLN.
14. Patients with a French social security in compliance with the French law relating to biomedical research (Article L.1121-11 of French Public Health Code).

Exclusion Criteria:

1. Rectal tumors (up to 15 cm from the anus)
2. Any metastasis.
3. Performance status ECOG ≥ 3.
4. Physical status score ASA ≥ 3.
5. Impaired cardiac function including any one of the following:

   5.1. LVEF < 45% or below the institutional lower limit of the normal range (whichever is higher) as determined by locally read echocardiogram. 5.2. Inability to determine the QT interval on ECG. 5.3. Complete left bundle branch block. 5.4. Use of a ventricular-paced pacemaker. 5.5. Congenital long QT syndrome or a known family history of long QT syndrome. 5.6. History of or presence of clinically significant ventricular or atrial tachyarrhythmias. 5.7. Clinically significant resting bradycardia (< 50 beats per minute). 5.8. QTc > 450 msec on the average of three serial baseline ECG (using the QTcF formula) as determined by central reading. If QTcF > 450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient rescreened for QTc. 5.9. History of clinically documented myocardial infarction. 5.10. History of unstable angina (during the last 12 months). 5.11. Other clinically significant heart disease (e.g. congestive heart failure or uncontrolled hypertension).
6. Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection).
7. History of significant congenital or acquired bleeding disorder unrelated to cancer.
8. Major surgery within 4 weeks prior to Day 1 of study or who have not recovered from prior surgery.
9. History of non-compliance to medical regimens or inability to grant consent.
10. Use of therapeutic coumarin derivatives (i.e., warfarin, acenocoumarol, phenprocoumon).
11. Patients actively receiving therapy with strong CYP3A4 inhibitors (e.g., erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil) and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
12. Patients actively receiving therapy with strong CYP3A4 inducers (e.g., dexamthasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbitol, St. John's Wort) and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
13. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery).
14. History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis.
15. Acute or chronic liver, pancreatic or severe renal disease considered unrelated to disease.
16. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
17. Patients who are: (a) pregnant, (b) breast feeding, (c) of childbearing potential without a negative pregnancy test prior to baseline and (d) female of childbearing potential unwilling to use contraceptive precautions throughout the trial and until two weeks after the end of treatment (post-menopausal women must be amenorrheic for at least 12 months to be considered of nonchildbearing potential). Contra-indication to nilotinib administration.
18. Previous or current malignancies other than colon cancer within the last 5 years, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin.
19. Emergency surgeries, including occlusion.
20. Previous enrolment in the present study.
21. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
ZAK expression level by immunohistochemistry on frozen material (surgical specimen) by Western blot and on paraffinembedded tissues section using an immunohistochemistry approach | Day 0
ZAK expression level by immunohistochemistry on frozen material (surgical specimen) by Western blot and on paraffinembedded tissues section using an immunohistochemistry approach | Day 7

SECONDARY OUTCOMES:
Efficacy of the 7day nilotinib treatment based on histological response as measured with tumour regression grade | Day 7
Efficacy of the 7day nilotinib treatment based on histological response as measured with the proportion of tumour necrosis | Day 7
Efficacy of the 7day nilotinib treatment based on histological response as measured with the type of tumour necrosis | Day 7
Incidence of Treatment Emergent Adverse Events as assessed by CTCAE v4.0 as assessed by CTCAE v4.0 | through study completion, an average of 2 years
Postoperative complications as assessed by Dindo and Clavien classification | through study completion, an average of 2 years
Maximum Plasma Concentration [Cmax] of nilotinib . | Day 7, day 8
Half-life of nilotinib | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No